CLINICAL TRIAL: NCT05087901
Title: Multifocal Electroretinography Before and After Silicone Oil Removal
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mohamed Abdel Hamid, Dr, Minia University
Other Study IDs: 34:3/2021
Record Dates: First submitted 2021-10-09; First posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Silicone Oil Filled Eyes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Silicone-filled eyes
  Interventions: Diagnostic Test: Multifocal electroretinogram

INTERVENTIONS:
Diagnostic Test: Multifocal electroretinogram — A device that records electric potentials generated by the retinal photoreceptors and neural elements in a multifocal fashion

SUMMARY:
This is a prospective observational study to investigate the changes in multifocal electroretinogram signal before and after silicone oil removal in silicone-filled eyes.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older who underwent pars plana vitrectomy for the repair of rhegmatogenous retinal detachment (RRD) and received silicone oil as an intraocular tamponade.

Exclusion Criteria:

* Patients will be excluded if they have a significant corneal opacity, uncontrolled intraocular pressure, a confounding macular pathology or optic nerve pathology or if silicone oil has been in the eye for longer than 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 30 patients will be recruited. We will include patients 18 years of age or older who underwent PPV for the repair of rhegmatogenous retinal detachment (RRD) and received silicone oil as an intraocular tamponade. Patients will be excluded if they have a significant corneal opacity, uncontrolled intraocular pressure, a confounding macular pathology or optic nerve pathology or if silicone oil has been in the eye for longer than 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Amplitude | Preoperative and 1 month postoperative recordings
  Change in amplitudes of P1 and N1 waves before and after silicone oil removal

CONTACTS AND LOCATIONS:
Locations (1):
- Minia University Hospital, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided